CLINICAL TRIAL: NCT01731236
Title: CARNIVAL Study: Gut Flora Dependent Metabolism of Dietary CARNItine and Phosphatidylcholine and cardioVAscuLar Disease
Acronym: CARNIVAL
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Stanley L Hazen, MD, PhD, Primary Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-544
Record Dates: First submitted 2012-01-23; First posted 2012-11-21 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Dietary Modification
Keywords: carnitine metabolism; gut flora; phosphatidylcholine
MeSH Terms: interventions — Carnitine; Choline; Anti-Bacterial Agents; Ciprofloxacin; Metronidazole; Vancomycin; Neomycin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Carnitine (No antibiotics, No aspirin) (Active Comparator): L-Carnitine 500 mg capsule by mouth, twice daily for 2 months. No aspirin for 1 month prior to starting study and remains off aspirin during study.
  Interventions: Dietary Supplement: Carnitine
- Choline (No Antibiotics, No aspirin) (Active Comparator): Choline 500 mg capsule by mouth, twice daily for 2 months. No aspirin for 1 month prior to starting study and remains off aspirin during study.
  Interventions: Dietary Supplement: Choline
- Antibiotics (Active Comparator): Antibiotics (Ciprofloxacin, Vancomycin, Metronidazole and Neomycin) Drug: Ciprofloxacin 500 mg, po, twice daily for 7 days (Other Names: Cipro)
  Drug: Metronidazole 500 mg, po, twice daily for 7 days (Other Names: Flagyl, Noritate, Rosadan, Vandazole, Flagyl ER, Vitazol)
  Drug: Vancomycin 125 mg, po, 4 times daily for 7 days (Other Names: Vancocin, Vancocin HCl, Pulvules, Vancoled, Novaplus, PremierPro Rx, Vancomycin HCl)
  Drug: Neomycin 1 gram, po, four times daily for 7 days (Other Names: Aminoglycoside)
  Interventions: Drug: Antibiotics
- Choline and Aspirin (Active Comparator): Choline supplement 500 mg capsule by mouth, twice daily for 2 months Drug: aspirin 81 mg by mouth, daily for 3 months (on aspirin for 1 month prior to starting study and 2 months with Choline supplementation during study)
  Other Names:
  Ecotrin, Bufferin, Ascriptin, Fasprin, Norwich Aspirin, Durlaza, Bayer Genuine Aspirin, Genacote, Bayer, Halfprin, Aspirtab, Aspir Low, Aspir-Trin
  Interventions: Drug: Choline and Aspirin
- Carnitine and Aspirin (Active Comparator): Carnitine supplement 500 mg capsule by mouth, twice daily for 2 months Drug: aspirin 81 mg by mouth, daily for 3 months (on aspirin for 1 month prior to starting study and 2 months with Carnitine supplementation during study)
  Other Names:
  Ecotrin, Bufferin, Ascriptin, Fasprin, Norwich Aspirin, Durlaza, Bayer Genuine Aspirin, Genacote, Bayer, Halfprin, Aspirtab, Aspir Low, Aspir-Trin
  Interventions: Drug: Carnitine and Aspirin

INTERVENTIONS:
Dietary Supplement: Carnitine — Group 1: Carnitine supplement for 2 months, No antibiotics, no aspirin for 3 months (1 month prior and during study)
  Arms: Carnitine (No antibiotics, No aspirin)
Dietary Supplement: Choline — Group 2: Choline supplement for 2 months, No antibiotics, no aspirin for 3 months (1 month prior and during study)
  Arms: Choline (No Antibiotics, No aspirin)
Drug: Antibiotics — Group 3: Carnitine or Choline for 2 months, antibiotic cocktail (Ciprofloxacin, Flagyl, Vancomycin, and Neomycin) for 1 week
  Other Names: Ciprofloxacin, Flagyl, Vancomycin, and Neomycin
  Arms: Antibiotics
Drug: Choline and Aspirin — Group 4: Choline supplement for 2 months plus aspirin 81 mg for 3 months (1 month prior to starting the study and 2 months during the study).
  Other Names: aspirin
  Arms: Choline and Aspirin
Drug: Carnitine and Aspirin — Group 5: Carnitine supplement for 2 months plus aspirin 81 mg for 3 months (1 month prior to starting the study and 2 months during the study).
  Other Names: aspirin
  Arms: Carnitine and Aspirin

SUMMARY:
The principal goal for the study is to examine the role gut flora plays in modulating metabolism of dietary carnitine and choline in humans.

DETAILED DESCRIPTION:
The principal goal for the study is to examine the role gut flora plays in modulating metabolism of dietary trimethylamine nutrients in humans. We have recently shown that dietary intake of two trimethylamines abundant in animal products, carnitine and the choline group of phosphatidylcholine (PC), are mechanistically linked to cardiovascular disease risk. We wish to further explore the metabolism of these nutrients in humans, and to test the hypothesis that the intestinal micro flora (gut flora) plays a critical role in generation of metabolites from dietary carnitine and choline/PC linked to cardiometabolic disease. We further hypothesize that the production of specific metabolites of carnitine and choline/PC are influenced by the composition of gut flora, and these may be altered by the preceding dietary patterns of the subjects. We therefore wish to test whether dietary supplementation with carnitine and/or choline alters the metabolism of carnitine and choline/PC in subjects. We also hypothesize that transient suppression or modulation of gut flora via short-term broad spectrum antibiotic therapy, or by reconstitution of micro flora composition via probiotic therapy, in healthy subjects, can alter the metabolism of carnitine and choline/PC. We will also examine the impact of low dose aspirin on these pathways by examining subjects before versus after taking aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or above.
* Able to provide informed consent and comply with study protocol

Exclusion Criteria:

* Significant chronic illness or end-organ dysfunction, including known history of heart failure, renal failure, pulmonary disease, hematologic diseases or pregnancy.
* Active infection or received antibiotics within 2 months of study enrollment
* Use of Over-The-Counter (OTC) probiotic within past 2 months, or ingestion of yogurt within past 7 days
* Chronic gastrointestinal disorders, or intolerance to probiotic therapy
* Having undergone Bariatric procedures or surgeries such as gastric banding or bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | December 2017
  Plasma levels of carnitine and multiple gut flora metabolites

SECONDARY OUTCOMES:
Secondary Outcome Measures | December 2017
  Alterations in plasma levels of cardio-metabolic risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L Hazen, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koeth RA, Lam-Galvez BR, Kirsop J, Wang Z, Levison BS, Gu X, Copeland MF, Bartlett D, Cody DB, Dai HJ, Culley MK, Li XS, Fu X, Wu Y, Li L, DiDonato JA, Tang WHW, Garcia-Garcia JC, Hazen SL. l-Carnitine in omnivorous diets induces an atherogenic gut microbial pathway in humans. J Clin Invest. 2019 Jan 2;129(1):373-387. doi: 10.1172/JCI94601. Epub 2018 Dec 10. PMID 30530985